CLINICAL TRIAL: NCT00039416
Title: A Phase II Study Of Gleevec (Imatinib Mesylate Formerly Known as STI-571) In Patients With Myelofibrosis
Brief Title: Imatinib Mesylate in Treating Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02895; NCI-2012-02895 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000069381; 11498A (Other: University of Chicago); 5669 (Other: CTEP); N01CM62201 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Myelomonocytic Leukemia; Essential Thrombocythemia; Polycythemia Vera; Primary Myelofibrosis
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Primary Myelofibrosis | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate once or twice daily on days 1-28. Courses repeat every 28 days for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have myelofibrosis. Imatinib mesylate may stop the growth of myelofibrosis by blocking certain enzymes necessary for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate (complete and partial) to STI-571 in patients with myelofibrosis.

II. To determine the safety of STI-571 in patients with myelofibrosis.

SECONDARY OBJECTIVES:

I. To determine the effects of STI-571 on bone marrow morphology (including effects on marrow fibrosis, osteosclerosis and cellularity) in patients with myelofibrosis.

II. To assess the effects of STI-571 on surrogate biologic endpoints including PDGFR expression (by immunohistochemistry), PDGFR signaling, and circulating progenitor (CD34 positive) cells.

III. To determine the effects of STI-571 on bone marrow cytogenetics in patients with an abnormal karyotype.

OUTLINE: This is a multicenter study. Patients are stratified according to Dupriez risk score (low vs intermediate vs high).

Patients receive oral imatinib mesylate once or twice daily on days 1-28. Courses repeat every 28 days for 12 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic confirmation of one of the following diseases-

  * Myeloid metaplasia with myelofibrosis (this includes all subtypes- chronic idiopathic myelofibrosis or agnogenic myeloid metaplasia, post thrombocythemic and post polycythemic myelofibrosis) or
  * Chronic myelomonocytic leukemia (CMMOL) with t(5;12)(q31-33;p12) or TEL-PDGFRβ rearrangement; patients with CMMOL and the t(5;7)(q31-33;q11.2) or other chromosomal translocations resulting in activation of PDGFR will also be eligible
  * Patients must have anemia (hemoglobin < 11 g/dL) or palpable splenomegaly (measured in cm from costal margin- to eligible); patients with palpable splenomegaly must have spleen size documented ultrasonographically as well; they must also meet standard diagnostic criteria for MMM* or CMMOL; patients with MMM must have thrombocytopenia (platelet count < 100 x 10^9/L) to be eligible; they must be Philadelphia chromosome or (BCR/ABL) rearrangement negative
  * Patients with CMMOL must also have the t(5;12)(q31-33;p12) or TEL-PDGFRβ rearrangement to be eligible
* The Italian diagnostic criteria for MMM

  * Necessary criteria

    * Diffuse bone marrow fibrosis
    * Absence of the Philadelphia chromosome or BCR-ABL rearrangement in peripheral blood cells
  * Optional criteria

    * Splenomegaly of any grade
    * Anisopoikilocytosis with tear drop erythrocytes
    * Presence of circulating immature myeloid cells
    * Presence of circulating erythroblasts
    * Presence of clusters of megakaryoblasts and anomalous megakaryocytes in bone marrow sections
    * Myeloid metaplasia
  * Diagnosis of MMM is acceptable if the following combinations are present

    * The two necessary criteria plus any other two optional criteria when splenomegaly is present OR
    * The two necessary criteria plus any other four optional criteria when splenomegaly is absent
* Patients may have had prior chemotherapy or radiation therapy including splenic irradiation; prior therapy with erythropoietin, GCSF or androgenic steroids is also permitted; there is no limit to number of prior regimens received; at least 4 weeks must have elapsed since prior chemo, radiation or other therapy
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Total bilirubin < 1.5 X institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal unless due to disease
* Serum creatinine < 2 X institutional upper limit of normal
* Patients must not be pregnant or nursing because STI-571 at the recommended therapeutic dose may be harmful to the developing fetus or newborn; for this reason women of child-bearing potential and men must agree to use an effective contraceptive method; women of reproductive potential must have a negative pregnancy test within 7 days prior to registration; since interactions with oral contraceptives cannot be excluded at present, male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug
* Ability to understand and the willingness to sign a written informed consent document
* World Health Organization (WHO) diagnostic criteria for CMMOL:

  * Persistent peripheral blood monocytosis > 1 x 10^9/L
  * Absence of the Philadelphia chromosome or BCR/ABL fusion gene
  * Fewer than 20% blasts in the blood or bone marrow
  * Dysplasia in one or more myeloid lineages; if myelodysplasia is absent or minimal, the diagnosis of CMML may still be made if the other criteria (1-3) are met and:

    * An acquired clonal cytogenetic abnormality is present in the marrow cells
    * The monocytosis has been persistent for at least 3 months
    * Other causes for monocytosis have been excluded

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to STI-571
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because STI-571 is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with STI-571, STI-571 should not be administered patients who are breastfeeding
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with STI-571; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Because warfarin is metabolized through the CYP450 system, and since gastrointestinal bleeding may occur with STI-571, no therapeutic anticoagulation with warfarin will be permitted in patients participating in this study; as an alternative, therapeutic anticoagulation may be accomplished using low-molecular weight heparin (e.g. Lovenox) or heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-04; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Clinical responses in terms of improvement in anemia and splenomegaly as previously published for myelofibrosis | Up to 12 months
Frequency of adverse events graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to 12 months
  Exact 95% confidence intervals generated using the binomial distribution.

SECONDARY OUTCOMES:
Progression-free survival | Up to 12 months
  Analyzed using the Kaplan-Meier method.
Bone marrow response | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Olatoyosi Odenike, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States